CLINICAL TRIAL: NCT01427257
Title: Phase 1 Open-Label Two-Way Cross Over Study to Assess the Pharmacokinetic Profile of Two Formulations of PB1023 Injection Following a Single Dose Administered By Subcutaneous Injection in Adult Subjects With Type 2 Diabetes Mellitus (T2DM)
Brief Title: Pharmacokinetic Profile of Two Formulations of PB1023 Following Single Subcutaneous Injection in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: PhaseBio Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PB1023-PT-CL-0002
Record Dates: First submitted 2011-08-29; First posted 2011-09-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PB1023 Formulation A (Active Comparator)
  Interventions: Drug: Single Dose PB1023
- PB1023 Formulation B (Active Comparator)
  Interventions: Drug: Single Dose PB1023
- PB1023 Formulation B (2-8C) (Active Comparator)
  Interventions: Drug: Single Dose PB1023

INTERVENTIONS:
Drug: Single Dose PB1023 — Single Dose PB1023 Formulation A
  Arms: PB1023 Formulation A
Drug: Single Dose PB1023 — Single Dose PB1023 Formulation B
  Arms: PB1023 Formulation B
Drug: Single Dose PB1023 — Single Dose PB1023 Formulation B
  Arms: PB1023 Formulation B (2-8C)

SUMMARY:
Primary objective:

To compare the pharmacokinetic profile of PB1023 after a single dose administered by subcutaneous injection of two formulations (concentrations).

Secondary objectives:

To evaluate the safety and tolerability of two formulations of PB1023 Injection administered as a subcutaneous injection in adult subjects with T2DM.

To evaluate the impact on the pharmacokinetic profile of PB1023 after a single 90 mg dose of formulation B (100 mg/mL) administered cold at 2 to 8°C by subcutaneous injection.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to sign a written informed consent and follow all study related procedures.
* Males or post menopausal or surgically sterile females age 18 - 75 years of age inclusive.
* Diagnosed with T2DM for ≥ 6 months.
* HbA1c of ≥ 6.0% if diet and exercise controlled, or ≥5.8% if taking one or more glucose lowering agents
* Weight ≥ 45 kg and BMI ≤ 40 kg/m2
* In otherwise stable health except for T2DM (no clinically significant laboratory abnormalities, vital signs, ECG findings or clinically significant underlying disease that would put the subject at risk for participation in the study).
* Receiving stable doses of concomitant medications for 30 days prior to dosing.
* Criteria for Participation in Period 3 only: Received PB1023 Injection at 50 mg/mL and 100 mg/mL during Period 1 or 2 of the study and had adequate pharmacokinetic samples collected for evaluation of their pharmacokinetic profile.

Exclusion Criteria:

* Currently taking Byetta® or Victoza®.
* Previously received PB1023 Injection other than under this study protocol.
* Known allergy or serious adverse effect to an approved or investigational GLP-1 receptor analog/agonist.
* Unstable cardiovascular disease defined as:

  * History of stroke, transient ischemic attack, or myocardial infarction within 6 months prior to the Screening visit.
  * Screening (duplicate supine reading) BP ≥ 160 mmHg (systolic) or ≥ 100 mmHg (diastolic).
  * Mean triplicate 12-lead ECG demonstrating QT interval (corrected) (QTc) > 450 msec in males and > 470 msec in females at the Screening visit, or a history or evidence of long QT syndrome.
* Based on contraindications/warnings identified with other GLP-1 receptor agonists, subjects will be excluded if they have:

  * History, symptoms or signs of pancreatitis or severe gastrointestinal disease (i.e., gastroparesis)
  * Personal or family history of medullary thyroid tumors or history of Multiple Endocrine Neoplasia Syndrome Type 2. Note: Abnormal serum calcitonin at screening will exclude the subject from participation.
* Clinically significant renal and/or hepatic dysfunction at screening as indicated by the following:

  * eGFR as calculated by MDRD of < 60 mL/min
  * Urine dipstick protein > 2+ (100 mg/dL) or urine protein 2+ and a Urine Protein/Creatinine ratio > 1.0 (> 1000 mg/g)
  * Alanine aminotransferase (ALT) > 2 x ULN
  * Aspartate aminotransferase (AST) > 2 x ULN
  * Serum bilirubin ≥ 1.6 mg/dL
* Pregnant or lactating females
* Known history of or active alcohol or drug abuse within 12 months prior to Screening or positive alcohol and/or drug screen.
* Positive for Human Immunodeficiency Virus (HIV) antibodies, Hepatitis B surface antigen (HBsAg) or Hepatitis C Virus (HCV) antibodies.
* Participating in any other study and have received any other investigational drug or device within 30 days prior to the Screening visit or are taking part in a non-drug study which in the opinion of the Investigator would interfere with the outcome of the study.
* Other medical (i.e., acute or chronic illness) or psychiatric condition which in the opinion of the Investigator would place the subject at increased risk, confound the primary study endpoint, or would preclude obtaining voluntary consent.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-02; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics | For each dosing period: Pre-dose, 1, 4, 8, 12 hours, 1, 2, 3, 4, 7 and 10 days post-dose
  The pharmacokinetic profile of two formulations of PB1023 will be compared. The following parameters will be evaluated: t1/2, AUC(inf), AUC(0-t), Tmax, Cmax, Elimination Rate Constant, Clearance and Distribution.

SECONDARY OUTCOMES:
Safety/Tolerability | 42 Days
  Safety will be evaluated by analyses of incidence of adverse events of interest (possibly related to the class of drug) and other adverse events. Vital signs, ECGs and safety laboratory parameters will also be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Matson, M.D., Principal Investigator — Prism Research
Locations (1):
- Prism Research, Saint Paul, Minnesota, United States